CLINICAL TRIAL: NCT07317258
Title: Evaluation of Cerebral Perfusion in Supine and Steep Trendelenburg Positions During Robotic Prostatectomy
Status: Not yet recruiting | Type: Observational
Sponsor: Hanife Kabukcu (Other)
Responsible Party: Sponsor-Investigator, Hanife Kabukcu, Prof. Dr., Akdeniz University
Organization: Akdeniz University (Other)
Other Study IDs: Cerebral Perfusion in Position
Record Dates: First submitted 2025-11-17; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-11

CONDITIONS: Cerebral Perfusion Pressure; Trendelenburg
Keywords: TRANSCRANİAL DOPPLER USG; CEREBRAL PERFUSİON; TRENDELENBURG; NIRS; EEG; PATİENT STATE İNDEKS; ROBOTİC SURGERY; PROSTATEKTOMİ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients Robotic Prostate Surgery: Men aged 18 to 80 undergoing robotic prostate surgery

SUMMARY:
Evaluation of Cerebral Perfusion in Supine and Steep Trendelenburg Positions During Robotic Prostatectomy Robotic endoscopic radical prostatectomy requires pneumoperitoneum and the steep Trendelenburg position to ensure optimal surgical visualization. However, this combination may increase intracranial pressure (ICP) and alter cerebral blood flow and oxygenation.

This study aimed to evaluate cerebral perfusion changes in patients undergoing robotic prostatectomy by using Transcranial Doppler (TCD) and Near-Infrared Spectroscopy (NIRS). Cerebral blood flow velocity in the middle cerebral artery and pulsatility index (PI) were measured to estimate ICP, while NIRS was used to assess cerebral oxygen saturation.

Additionally, arterial blood gas parameters (PCO₂, PO₂, Hb), end-tidal CO₂, and mean arterial pressure (MAP) were recorded. Pre- and postoperative Mini-Mental State Examination (MMSE) scores were compared to evaluate potential cognitive effects.

The aim was to determine the relationship between ICP estimation, cerebral oxygenation, and hemodynamic variables during supine and steep Trendelenburg positions in robotic prostatectomy.

DETAILED DESCRIPTION:
The use of robotic endoscopic radical prostatectomy has the potential to improve surgical outcomes and reduce complications compared to open radical prostatectomy. Robotic endoscopic abdominal surgery involves carbon dioxide (CO₂) insufflation to create pneumoperitoneum and requires the Trendelenburg position to provide adequate surgical visualization.

An increase in intra-abdominal pressure due to pneumoperitoneum leads to various physiological changes. The combination of steep Trendelenburg positioning and pneumoperitoneum during robotic prostatectomy is known to cause intracranial hypertension. The elevation of intra-abdominal pressure and Trendelenburg positioning increases intracranial pressure (ICP) and alters cerebral blood flow (CBF). These changes in cerebral hemodynamics may have detrimental effects on cerebral oxygenation.

Several invasive and non-invasive techniques are available for monitoring ICP and cerebral perfusion pressure (CPP). Among non-invasive methods, Transcranial Doppler ultrasonography (TCD) and Near-Infrared Spectroscopy (NIRS) are reliable and safe monitoring tools.

TCD measures blood flow velocities in the major arteries of the Circle of Willis. Based on TCD-derived data, several formulas have been proposed to estimate ICP, such as the Pulsatility Index (PI) and Resistance Index (RI).

PI is calculated using the formula:

PI = (Peak systolic velocity - End diastolic velocity) / Mean velocity. A normal PI typically ranges between 0.5 and 1.2. Under normal systemic hemodynamic conditions, an elevated PI (particularly >2) suggests reduced cerebral perfusion pressure (CPP).

RI is calculated as:

RI = (Peak systolic velocity - End diastolic velocity) / Peak systolic velocity.

An RI greater than 0.75-0.8 is considered abnormal. RI is conceptually similar to PI (both increase in cases of low CPP), although PI is more widely used in clinical practice.

Normal ICP values vary with age and body position, but are generally 5-15 mmHg in healthy supine adults, 3-7 mmHg in children, and 1.5-6 mmHg in infants.

In cases of elevated ICP or circulatory hypotension, cerebral perfusion pressure (CPP) decreases. CPP is calculated as the difference between mean arterial pressure (MAP) and ICP. MAP is obtained by adding one-third of the pulse pressure (the difference between systolic and diastolic pressure) to the diastolic pressure.

NIRS technology was recently developed to enable continuous and non-invasive monitoring of regional cerebral tissue oxygen saturation for various clinical indications. The differing absorption spectra of oxygenated and deoxygenated hemoglobin at different light wavelengths allow for assessment of the balance between cerebral oxygen supply and demand.

In this study, the correlation between cerebral oxygen saturation measured by NIRS and estimated ICP calculated from TCD-derived middle cerebral artery (MCA) flow velocity and pulsatility index was evaluated. In addition, arterial blood gas parameters (PCO₂, PO₂, hemoglobin), end-tidal CO₂ (EtCO₂), and mean arterial pressure (MAP) were included in the analysis.

Preoperative and postoperative Mini-Mental State Examination (MMSE) tests were administered to assess potential cognitive changes and to compare our non-invasive monitoring results with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

Male patients aged 18 to 80 years

ASA physical status I-III

Scheduled for robotic prostate surgery under general anesthesia

Able and willing to provide written informed consent

Exclusion Criteria:

Decline or inability to provide informed consent

Age <18 years or >80 years

Inability to perform ultrasonographic measurements or to maintain the required surgical position

Presence of intracranial space-occupying lesions

History of cerebrovascular accident (CVA) or carotid artery occlusion

Known neurological disorders (e.g., epilepsy)

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients aged 18 to 80 years undergoing robotic prostate surgery under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Cerebral Oxygenation Measured by Near-Infrared Spectroscopy (NIRS) | 1.Upon arrival in the operating room (baseline) 2.10 minutes after endotracheal intubation 3.30 minutes after placement in the Trendelenburg position 4.10 minutes before returning to the supine position 5. Postoperative 1 hour
  Cerebral oxygenation will be assessed using near-infrared spectroscopy (NIRS). Regional cerebral oxygen saturation (%) will be continuously monitored, and values will be recorded at predefined perioperative time points.
Middle Cerebral Artery Blood Flow Velocity Measured by Transcranial Doppler Ultrasonography (TCD) | 1.Supine position, 10 minutes after endotracheal intubation 2.30 minutes after placement in the Trendelenburg position 3.10 minutes before returning to the supine position 4.After returning to the supine position 5.Postoperative 1 hour
  Middle cerebral artery (MCA) blood flow velocity will be measured using transcranial Doppler ultrasonography (TCD). MCA mean flow velocity (cm/s) will be recorded at predefined perioperative time points.

SECONDARY OUTCOMES:
Mean Arterial Pressure (MAP) at Predefined Perioperative Time Points | 1.Upon arrival in the operating room 2.10 minutes after endotracheal intubation 3.30 minutes after placement in the Trendelenburg position 4.10 minutes before returning to supine 5.Postoperative 1 hour
  Mean arterial pressure (mmHg) will be recorded continuously and extracted at predefined perioperative time points to assess hemodynamic changes associated with patient positioning.
End-Tidal CO₂ (EtCO₂) at Predefined Perioperative Time Points | 1.Upon arrival in the operating room 2.10 minutes after endotracheal intubation 3.30 minutes after placement in the Trendelenburg position 4.10 minutes before returning to supine 5.Postoperative 1 hour
  End-tidal carbon dioxide (mmHg) will be monitored continuously and documented at several standardized perioperative time points to assess potential effects of Trendelenburg positioning and pneumoperitoneum on ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Hanife Kabukcu, Study Director — Akdeniz University; Sinem Omca, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
IPD used in publishing the results
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be available from October 5, 2025, to October 30, 2026, and will be shared after the study results have been finalized and published.
Access Criteria: finalization of the results

REFERENCES:
- [Result] Kalmar AF, Dewaele F, Foubert L, Hendrickx JF, Heeremans EH, Struys MM, Absalom A. Cerebral haemodynamic physiology during steep Trendelenburg position and CO(2) pneumoperitoneum. Br J Anaesth. 2012 Mar;108(3):478-84. doi: 10.1093/bja/aer448. Epub 2012 Jan 17. PMID 22258202
- [Result] Kalmar AF, Foubert L, Hendrickx JF, Mottrie A, Absalom A, Mortier EP, Struys MM. Influence of steep Trendelenburg position and CO(2) pneumoperitoneum on cardiovascular, cerebrovascular, and respiratory homeostasis during robotic prostatectomy. Br J Anaesth. 2010 Apr;104(4):433-9. doi: 10.1093/bja/aeq018. Epub 2010 Feb 18. PMID 20167583